CLINICAL TRIAL: NCT05427383
Title: A Randomized, Multicenter, Phase Ⅱ/Ш Clinical Study to Evaluate the Efficacy of KN026 in Combination With Chemotherapy in Subjects With HER2 Positive Advanced Unresectable or Metastatic Gastric Cancer (Including Gastro-esophageal Junction Adenocarcinoma) Who Have Failed First-line Therapy.
Brief Title: KN026 in Combination With Chemotherapy in HER2 Positive Gastric Cancer Subjects Who Have Failed First-line Therapy
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KN026-001
Record Dates: First submitted 2022-06-14; First posted 2022-06-22 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Stomach Cancer
Keywords: Stomach Neoplasm; Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — Paclitaxel; Docetaxel; Irinotecan

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KN026 + Paclitaxel/ Docetaxel/ Irinotecan (Experimental): IV KN026 at 30 mg/kg on D1 and IV Paclitaxel at 175 mg/m² on D1 or IV Docetaxel at 75 mg/m² on D1 or IV Irinotecan at 125 mg/m² on D1, D8, Q3W
  Interventions: Drug: KN026/Placbo Injection; Drug: Paclitaxel Injection; Drug: Docetaxel Injection; Drug: Irinotecan Injection
- Placebo + Paclitaxel/ Docetaxel/ Irinotecan (Experimental): IV Placebo at 30 mg/kg on D1 and IV Paclitaxel at 175 mg/m² on D1 or IV Docetaxel at 75 mg/m² on D1 or IV Irinotecan at 125 mg/m² on D1, D8, Q3W
  Interventions: Drug: KN026/Placbo Injection; Drug: Paclitaxel Injection; Drug: Docetaxel Injection; Drug: Irinotecan Injection

INTERVENTIONS:
Drug: KN026/Placbo Injection — IV KN026/Placebo at 30 mg/kg on D1, Q3W
Drug: Paclitaxel Injection — IV Paclitaxel at 175 mg/m² on D1, Q3W
Drug: Docetaxel Injection — IV Docetaxel at 75 mg/m² on D1, Q3W
Drug: Irinotecan Injection — IV Irinotecan at 125 mg/m² on D1, D8, Q3W

SUMMARY:
KN026-001 is a two-stage study (Open-label stage/Randomized stage). Open-label stage is designed to evaluate the safety and efficacy of KN026 and chemotherapy when given together. Randomized stage is designed to evaluate the OS and PFS in patients receiving KN026 and chemotherapy compared to patients receiving placebo and chemotherapy.

DETAILED DESCRIPTION:
KN026-001 is a two-stage randomized, multicenter, phase Ⅱ/Ⅲ clinical study to evaluate the efficacy of KN026 in combination with chemotherapy in subjects with HER2-positive advanced unresectable or metastatic gastric cancer, including adenocarcinoma of the gastro-esophageal junction, who have failed first-line therapy.

Stage 1 is an open-label, multicenter, phase Ⅱ study to evaluate the safety and ORR in subjects receiving KN026 in combination with chemotherapy. Stage 2 is a randomized, double-blind, placebo-controlled phase Ш study to evaluate the OS and PFS in subjects receiving KN026 in combination with chemotherapy compared to placebo in combination with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years;
2. Histologically or cytology-confirmed HER2-positive locally advanced, recurrent, or metastatic gastric cancer (including adenocarcinoma of the gastro-esophageal junction); HER2 positive is defined as IHC 3+, or IHC 2+ with ISH test positive (HER2/CEP17 ratio ≥ 2.0, or mean HER2 copy number ≥ 6.0 signals/cell);
3. Failure of at least first-line standard therapy (trastuzumab plus chemotherapy); Note: Neoadjuvant/adjuvant therapy previously administered with a trastuzumab-containing regimen can be considered first-line therapy if the subject has progressed disease during neoadjuvant/adjuvant therapy or within 6 months of completion of treatment;
4. Stage 1 : At least one measurable lesion at baseline according to RECIST 1.1; Stage 2: At least one evaluable lesion at baseline according to RECIST 1.1; the area must not have received previous radiotherapy, or there must be evidence of significant progression after the end of radiotherapy;
5. ECOG Performance Status of 0 to 1.
6. Life expectancy ≥ 3 months.
7. 7. The function of major organs must meet the following criteria : Hemoglobin (Hb) ≥ 90 g/L; Absolute neutrophil (ANC) ≥ 1.5×10^9/L; Platelet (PLT) ≥ 90×10^9/L; (No whole blood or component blood transfusion in the last 14 days; no pro-hematopoietic cytokines used in the last 7 days); AST, ALT ≤2.5× ULN (upper limit of normal value) (if liver metastases, AST, ALT ≤5×ULN); Total bilirubin (TBIL) ≤1.5×ULN; Albumin≥ 28 g/L; creatinine clearance ≥ 50 mL/min (standard Cockcroft-Gault formula applied); Activated partial thromboplastin time (APTT) ≤ 1.5×ULN, international normalized ratio (INR)/or prothrombin time (PT) ≤ 1.5×ULN; (It is allowed to receive anticoagulants at low stable doses, eg at a dose of aspirin 100 mg/day);
8. Left ventricular ejection fraction (LVEF) ≥ 50% or lower limit of normal (LLN) in local sites, measured by echocardiography (ECHO), cardiac radionuclide scanning (MUGA) only in the absence of ECHO, with consistency at baseline and follow-up measurements;
9. Subjects agreed to use effective contraception during the study and for 6 months after the last dose (women of childbearing age must confirm a negative serum pregnancy test within 7 days prior to enrollment);
10. Female and male patient of childbearing age must agree to take adequate contraceptive measures during the entire study period and through at least 6 months after the last dose of study drug. (Women of childbearing age must have a negative pregnancy test prior to study entry.)
11. Subjects are able and willing to comply with the study protocol.

Exclusion Criteria:

1. Subjects with untreated active brain metastases; Subjects will be admitted if their brain metastases have been treated and the metastases are stable (brain imaging at least 4 weeks prior to the first dose showed stable lesions with no new CNS symptoms, or CNS symptoms have returned to baseline and no hormonal therapy is required at least 14 days prior to the first dose of the investigational treatment), and there is no evidence of new or enlarged original brain metastases;
2. Other investigational medications received within 4 weeks prior to the first study treatment, based on the time of the last trial dose;
3. Antineoplastic therapy such as chemotherapy, small molecule inhibitors, immunotherapy (such as interleukin, interferon, or thymosin) within 4 weeks or 5 half-lives (whichever is shorter but at least 2 weeks) prior to the first study treatment; Have received Chinese herbal treatment with antitumor activity within 14 days before administration;
4. Subjects recieved major surgery (e.g., transabdominal, transthoracic, etc.) within 28 days prior to the first study treatment; does not include minor procedures such as diagnostic puncture or infusion device implantation), or major surgery is expected to be required during the study;
5. Previous cumulative doses of doxorubicin exceeding 320 mg/m^2, or equivalent conversion of other anthracyclines (anthracycline equivalent: 1 mg doxorubicin = 2 mg epirubicin = 2 mg pyrrubicin = 2 mg daunorubicin = 0.5 mg normethoxydaunorubicin = 0.45 mg mitoxantrone; except doxorubicin liposomes);
6. Previous use of anti-HER2 therapy other than trastuzumab (eg, ADC, dual-antibody, small molecule targeted therapy, etc.).
7. Pregnant or lactating women; or intend pregnancy during the trial or within 6 months of the end of the trial;
8. Subjects with a history of life-threatening allergies or known allergies to protein drugs or recombinant proteins or to one of excipients in KN026 drugs (histidine, glacial acetic acid, sucrose, and polysorbate 20) who have had a severe hypersensitivity reaction to trastuzumab.
9. Adverse events have not returned to CTCAE 5.0 grade ≤ grade 1 or baseline from previous anti-tumor treatments , except for alopecia, skin pigmentation and those assessed by the investigators without potential safety risk.
10. Uncontrollable diarrhoea (≥grade 2 that does not improve within 48 hours of medication);
11. Subjects with the following history of cardiovascular disease:

    * Subjects with uncontrolled hypertension (defined as sustained systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg despite antihypertensive medication);
    * Any history of symptomatic congestive heart failure (NYHA classification II-IV); the absolute value of LVEF decreased by ≥10% and absolute value < 50% , or the absolute value of LVEF decreased by ≥15% , during or after treatment with trastuzumab or other anti-HER2 treatment;
    * History of myocardial infarction within 6 months before treatment of the first dose;
    * Subjects with angina and unstable angina within three months prior to treatment in the first dose;
    * Severe arrhythmias and conduction abnormalities requiring antiarrhythmic therapy other than β-blockers or digoxin (except atrial fibrillation and paroxysmal supraventricular tachycardia) within 6 months prior to treatment in the first dose;
    * QTcF > 450 ms (male); QTcF > 470ms (Female);
    * Other heart diseases that the investigators consider clinically significant;
12. Poorly controlled systemic diseases judged by investigators, including diabetes;
13. Severe chronic or active infections requiring systemic antibacterial, antifungal, or antiviral therapy (eg, anti-infective drugs have been used for more than 1 week before the trial and will continue to be used), including tuberculosis infection;
14. Received systemic corticosteroids (> 10 mg/day of prednisone, or equivalent amounts of other corticosteroids) within 2 weeks prior to treatment in the first dose; inhaled steroids or topical cortisol is permitted, corticosteroids are allowed for pre-treatment of certain chemotherapy drugs, and short-term (≤ 7 days) are allowed for the prevention or treatment of contrast allergy;
15. History of noninfectious interstitial lung disease, or interstitial pneumonia requiring hormonal therapy;
16. History of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency disease, or a history of organ transplantation;
17. Active HBV [HBsAg or HBcAb-positive with HBV DNA > 500 IU/mL (or 2500 copies/mL)] or HCV infection [subjetcs with polymerase chain reaction (PCR)-negative HCV ribonucleic acid (RNA) can participate in this study] or HIV-positive or syphilis antibody positive (confirmed);
18. History of any other malignant tumors within five years prior to the first dose, except cured cutaneous squamous cell carcinoma, basal cell carcinoma, non-muscle-invasive bladder cancer, localized low-risk prostate cancer [defined as stage ≤ T2a, Gleason score ≤ 6, and PSA ≤ 10 ng/mL at prostate cancer diagnosis (if measured) who have received radical therapy and no biochemical recurrence of prostate-specific antigen (PSA) can participate in this study], cervical/breast cancer in situ who have received radical treatment without any signs of recurrence and metastasis;
19. Cavity effusion (pleural effusion, ascites, pericardial effusion, etc.) requiring drainage or diuretic therapy, within 2 weeks prior to the first dose of treatment; Diuretics for other reasons are permitted;
20. Known mismatch repair deficient (dMMR) or highly unstable microsatellite (MSI-H) without previous PD-1/PD-L1 monoclonal antibody therapy;
21. Unintentional weight loss of ≥5% within 1 month prior to the first dose, despite peripheral or central venous nutritional support;
22. Inability to tolerate or refuse chemotherapy required by the protocol;
23. The investigator considered the subject to be unsuitable for participation in this clinical study due to the presence of any clinical or laboratory abnormalities or history of systemic disease or other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) according to RECIST 1.1 by IRC | Up to 2.5 years
  The time from the first dose of study treatment to the date of documented disease
Overall Survival (OS) according to RECIST 1.1 by IRC | Up to 2.5 years
  The time from the first dose of study treatment until the date of death from any cause

SECONDARY OUTCOMES:
ORR according to RECIST 1.1 by Investigator's Assessment and IRC | Up to 2.5 years
  The percentage of patients with a complete response (CR) or partial response (PR)
DCR according to RECIST 1.1 by Investigator's Assessment and IRC | Up to 2.5 years
  Number of subjects who achieved a best response of CR, PR, or SD during treatment
DOR according to RECIST 1.1 by Investigator's Assessment and IRC | Up to 2.5 years
  The time from the first objective response (CR or PR) to documented PD, clinical progression, or death from any cause
Progression Free Survival (PFS) according to RECIST 1.1 by Investigator's Assessment | Up to 2.5 years
  The time from the first dose of study treatment to the date of documented disease
Frequency and Severity of Adverse Events according to NCI CTCAE 5.0 | Up to 2.5 years
  Number of participants with treatment-related adverse events as assessed by CTCAE 5.0
The concentration of KN026 drug in serum | Up to 2.5 years
  The concentration of KN026 drug in serum
Incidence and titer of anti-drug antibody (ADA) | Up to 2.5 years
  Incidence and titer of anti-drug antibody (ADA)
Incidence of neutralizing Antibody，Nab | Up to 2.5 years
  Incidence of neutralizing Antibody，Nab

OTHER OUTCOMES:
To explore the correlation of gene mutation status and the efficacy | Up to 2.5 years
  Exploration of drug resistance mechanism , Explore predictive biomarkers
Subjects will be assessed using the European Quality of Life 5 Dimensions and 5 Lines (EQ-5D-5L) scales | Up to 2.5 years
  It is a vertical visual analogue scale that takes values between 100 (best imaginable health) and 0 (worst imaginable health), on which patients provide a global assessment of their health.
Subjects will be assessed using the Quality of Life Questionnaire-Core 30 (QLQ-C30) scales | Up to 2.5 years
  The QLQ-C30 is composed of six functioning scales (including a measure for global quality of life), three symptom scales, and six single items. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Subjects will be assessed using the Quality-of-life Questionnaire Oesophago Gastric module 25 (EORTC QLQ OG25) scales | Up to 2.5 years
  Quality-of-life Questionnaire Oesophago Gastric module 25 (EORTC QLQ OG25): Description: All of the scales and single-item measures range in score from 0 to 100. A high score for all the scales and single-items represents a high level of symptomatology or problems.
Change from baseline in CEA (carcinoembryonic antigen) | Up to 2.5 years
Change from baseline in CA19-9 (carbohydrate antigen 199) | Up to 2.5 years
Change from baseline in CA72-4 (carbohydrate antigen 724) | Up to 2.5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided